CLINICAL TRIAL: NCT01938066
Title: Clinical Outcomes for Patients With Acute Surgical Wounds Treated With Procellera and Negative Pressure Therapy Versus Standard of Care, Negative Pressure Therapy Only
Brief Title: Procellera and Negative Pressure Therapy for Acute Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gayle Gordillo (Other)
Collaborators: Vomaris Innovations (Industry)
Responsible Party: Sponsor-Investigator, Gayle Gordillo, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013H0028
Record Dates: First submitted 2013-09-04; First posted 2013-09-10 (Estimated); Results first posted 2016-04-21 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Wound
Keywords: procellera
MeSH Terms: conditions — Wounds and Injuries | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Negative Pressure with Procellera (Active Comparator): Arm 2 is Negative Pressure Therapy and Procellera Dressing under the sponge dressing of the Negative Pressure Therapy. The dressing will be changed at the end of 5 days. This is the intervention arm of the study.
  Interventions: Device: Procellera; Device: negative pressure therapy
- Negative Pressure Therapy only (Sham Comparator): Arm 1 is Negative Pressure Therapy only with no Procellera Dressing and the dressing is changed every other day per standard of care when you use Negative Pressure Therapy with no dressing underneath the sponge.
  Interventions: Device: negative pressure therapy

INTERVENTIONS:
Device: Procellera — bioelectric wound dressing
  Arms: Negative Pressure with Procellera
Device: negative pressure therapy

SUMMARY:
The purpose of this study is to determine if Procellera speeds wound healing. The study will examine colonization (bacterial growth), pain and pain medication and reduced cost of care by using Procellera (an antimicrobial agent) under Negative Pressure Therapy placed on the wound after abdominal wall surgery. Procellera is a single layer dressing that helps to kill germs that cause infections. Negative Pressure Therapy is a vacuum device with a sponge that is placed in your wound to help heal the wound faster.

DETAILED DESCRIPTION:
The study will consent 30 patients undergoing surgery through the abdominal wall and the skin incision will intentionally be left open. Subjects will be randomized using a random number generator. Each number will be placed in an envelope numbered 1-30. Arm 1 will be even numbers and Arm 2 will be odd numbers. A researcher not affiliated with the study will generate the numbers and place them in the envelopes. Arm 1 will place fifteen subjects on Negative Pressure Therapy Only and Arm 2 will place fifteen subjects on Negative Pressure and Procellera. Arm 1 (Negative Pressure Only) will have their dressing changed 3 times per week which is the standard of care for Negative Pressure Therapy. Arm 2 (Negative Pressure Therapy and Procellera) will have their dressing changed every 5 days. Arm 1 and 2 will have a tissue specimen taken on the 5th day only. The tissue will be taken from debrided material and sent for culture. The Negative Pressure Therapy Sponge, which is discarded after each dressing change, will be collected, lavaged with saline and the cells will be examined for macrophage function and the wound fluid will be tested for inflammation response. Photographs, wound measurements, pain scale and pain medication will also be completed at each dressing change. We will check the progress of the wound along with your surgeon during the subject's 30 day surgical follow up in the surgeon's office. The wound will be measured (if not healed), photograph's taken and their pain level assessed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old that are undergoing abdominal wall surgery

Exclusion Criteria:

* Below 18 years old and not having abdominal wall surgery

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gayle M Gordillo, MD, Principal Investigator — Ohio State University
Locations (1):
- University Hosptial East, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Negative Pressure With Procellera: Arm 2 is Negative Pressure Therapy and Procellera Dressing under the sponge dressing of the Negative Pressure Therapy. The dressing will be changed at the end of 5 days. This is the intervention arm of the study.
  Procellera: bioelectric wound dressing
  negative pressure therapy
- Negative Pressure Therapy Only: Arm 1 is Negative Pressure Therapy only with no Procellera Dressing and the dressing is changed every other day per standard of care when you use Negative Pressure Therapy with no dressing underneath the sponge.
  negative pressure therapy
Period: Overall Study
Arm/Group | Negative Pressure With Procellera | Negative Pressure Therapy Only
Started | 15 | 15
Completed | 14 | 13
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Negative Pressure With Procellera | Negative Pressure Therapy Only | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 14
  >=65 years | 3 | 10 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10) | 58.3 (12) | 56.8 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 8 | 12 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27
Weight [Mean (Standard Deviation); unit: lbs] | 215.5 (66.2) | 202.1 (85.1) | 210.6 (74.3)

OUTCOME MEASURES:

1. Primary Outcome: Wound Infection
Description: At the end of 5 days all subjects will get a Culture and Sensitivity to see if they have an infection or what type of infection they have in the wound
Time Frame: At the end of 5 days
Measure: Number; unit: participants
Arm/Group | Negative Pressure With Procellera | Negative Pressure Therapy Only
Number analyzed (Participants) | 13 | 12
participants | 13 | 12

2. Secondary Outcome: Amount of Pain Medication Used (Morphine)
Description: will measure the amount of pain medication used (morphine)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Negative Pressure With Procellera | Negative Pressure Therapy Only
Number analyzed (Participants) | 14 | 13
mg | 139.29 (116.05) | 178.55 (147.28)

ADVERSE EVENTS:
Description: The use of Procellera presented no risks during the study timeline. The subjects were not placed on Procellera if they have any sensitivity to zinc, silver or have uncontrolled bleeding.
Arm/Group | Negative Pressure With Procellera | Negative Pressure Therapy Only
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No